CLINICAL TRIAL: NCT02986789
Title: Evaluation of Impacts of Continuous Non-Invasive Intra-Operative Hemoglobin and PVI Monitoring on Intra-Operative and Post-Surgical Clinical Outcomes
Brief Title: Continuous Non-Invasive SpHb and PVI Monitoring on Intra-Operative and Post-Surgical Clinical Outcomes
Status: Terminated | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BIGT0001
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Results first posted 2022-01-05 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Unapproved Device: Yes

ARMS (2):
- Control Group (No Intervention): Clinicians will be performing blood transfusions using hospital standard of care procedures.
- Evaluation Group (Experimental): Clinicians will be guiding blood transfusions using SpHb with In vivo feature as a trigger for laboratory blood draws and PVi to inform fluid administration decisions in addition to hospital standard of care procedures.
  Interventions: Device: In vivo SpHb and PVi Monitoring

INTERVENTIONS:
Device: In vivo SpHb and PVi Monitoring — Pulse oximeter finger sensor that simultaneously monitors noninvasive hemoglobin (SpHb) and pleth variability index (PVi)
  Arms: Evaluation Group

SUMMARY:
The study evaluates the use of noninvasive hemoglobin with In Vivo feature and PVi monitoring using pulse-oximetry based technologies and their effect on the management of transfusion and infusion decisions and clinical outcomes for the surgical patient.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing major surgeries associated with possibility of significant blood loss (e.g. such that blood is cross-matched and available before the start of the case as per hospital routine practice) under general anesthesia.
* At least one finger available and accessible for performing non-invasive hemoglobin monitoring.

Exclusion Criteria:

* Patient has skin abnormalities affecting the digits such as psoriasis, eczema, angioma, scar tissue, burn, fungal infection, substantial skin breakdown, nail polish or acrylic nails that would prevent the proper fit and application of the sensors
* Procedures performed using robotics surgery
* Any patients with a known hemoglobinopathy
* Any patients undergoing Cardio-Pulmonary Bypass (CPB)
* Any patients who cannot be transfused or has refused consent for a blood transfusion
* Patients being treated by any artificial oxygen carriers within 30 days of hospital stay
* Patients being managed outside of an operating room in the participating centers, or in operating room with conditions not conducive to perform and complete the study procedures (including use of the hemoglobin monitoring device)
* Patients younger than 18 years old
* Patients who are pregnant
* Patients with cardiac arrhythmia
* Patients with tidal volume setting < 6ml/kg
* Patients with PEEP >= 10cm H2O
* Patients undergoing cardiac and/or any open chest procedures
* Emergency patients due to the foreseeable difficulty in consenting
* Patients deemed not suitable for study at the discretion of the Principal Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Evaluation Group
Started | 43 | 0
Completed | 43 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants enrolled in the evaluation group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Evaluation Group | Total
Number analyzed (Participants) | 43 | 0 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 0 | 29
  >=65 years | 14 | 0 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 0 | 22
  Male | 21 | 0 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 9 | 0 | 9
  Hispanic, Latino, or Spanish origin | 2 | 0 | 2
  White or Caucasian | 32 | 0 | 32
Region of Enrollment [Number; unit: participants]
  United States | 43 |  | 43

OUTCOME MEASURES:

1. Primary Outcome: Average Volume of Allogenic RBC Transfused Intra-operatively
Description: Reduction in overall allogenic transfusion is defined as the decrease in volume of transfusion of the intervention group relative to control group, intra-operatively.
Time Frame: Approximately 6-8 hours
Population: Only historical chart review was able to be completed for the 43 control subjects, therefore there are no results to report for the control group. This study was not able to meet the enrollment target for the control and intervention groups, and therefore average volume of allogenic RBC transfused intra-operatively could not be defined (primary outcome measures).
Arm/Group | Control Group | Evaluation Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: No participations were enrolled in the evaluation group.
Arm/Group | Control Group | Evaluation Group
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/0
Other Adverse Events (participants affected / at risk) | 0/43 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT02986789/Prot_SAP_000.pdf